CLINICAL TRIAL: NCT07210567
Title: Mindfulness-based Ecological Momentary Intervention for Smoking Cessation Among Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Min-Jeong Yang, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2024002019; R00CA271040 (NIH)
Record Dates: First submitted 2025-09-17; First posted 2025-10-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation
Keywords: quit smoking; cancer survivors
MeSH Terms: conditions — Smoking Cessation | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Participants will receive brief counseling, nicotine replacement therapy, and intervention content delivered via the app.
  Interventions: Behavioral: Mindfulness
- Quitline (Active Comparator): Participants will be referred to Quitline to receive standard care for smoking cessation.
  Interventions: Behavioral: Quitline

INTERVENTIONS:
Behavioral: Mindfulness — Participants will complete 4 counseling sessions (30 minutes), download and use a smartphone app for 4 weeks, complete 4 online surveys (baseline, quit date, end of treatment, and 3-month follow-up), and a brief phone call at the end of treatment to provide feedback. Participants will use the app every day to complete daily diaries and ecological momentary assessments (EMAs), receive brief mindful skills, and practice formal mindfulness meditations (5-30 minutes). Participants will also be provided with nicotine patches.
  Arms: Mindfulness
Behavioral: Quitline — Participants will be referred to Quitline to receive standard care smoking cessation treatment, including counseling and nicotine patches. Participants will complete 4 online surveys (baseline, quit date, end of treatment, and 3-month follow-up) and a brief phone call at the end of treatment to provide feedback. Participants will use the app every day to complete daily diaries.
  Arms: Quitline

SUMMARY:
The purpose of the study is to develop a new quit-smoking treatment among individuals with a cancer diagnosis using a smartphone app.

DETAILED DESCRIPTION:
The study aims to test the feasibility and acceptability of the smartphone app we developed in conjunction with face-to-face brief cessation counseling and nicotine replacement therapy in a two-arm randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* smoked ≥1 cigarette per day (even one or two puffs) within the past 30 days
* having been diagnosed with cancer
* being motivated to quit in the next 30 days
* having a valid home address and functioning phone number
* being able to read, write, and speak English
* having a smartphone that allows installation of the app
* willingness to download the app

Exclusion Criteria:

* being enrolled in a smoking cessation program
* current use of smoking cessation medications
* evidence of current psychosis
* current/planning pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
System Usablity Scale | End of Treatment at 4 Weeks
  Perceived usability and learnability of the app will be measured on a 5-point scale (1=strongly disagree; 5=strongly agree).
Client Satisfaction Questionnaire | End of Treatment at 4 Weeks
  Perceived satisfaction with the treatment will be assessed on a 4-point scale (1=very dissatisfied; 4=very satisfied).
Percentage of Participants That Completed Questionnaires | 3-month follow-up
  Completion of follow-up assessment will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Jeong Yang, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Institute for Nicotine & Tobacco Studies, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No